CLINICAL TRIAL: NCT04080479
Title: Bolus Versus Continuous Enteral Feeding in Critically Ill Patients
Brief Title: Bolus Versus Continuous Enteral Tube Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FNO-KARIM-12-Enteral_Feeding
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Trauma Injury; Major Abdominal Surgery; Sepsis
Keywords: bolus enteral feeding; continuous enteral feeding; protein synthesis; nutritional parameters
MeSH Terms: conditions — Accidental Injuries; Sepsis | interventions — Muscle Strength

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomized into one of the two study arms.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus enteral feeding (Experimental): The patients randomized into this study arm will receive bolus enteral feeding. The study subjects will undergo the following interventions:
  * Quadriceps Muscle Layer Fitness measurement
  * Muscle Strength measurement
  * Acute Physiology and Chronic Health Evaluation
  * Sequential Organ Failure Assessment
  * Nutritional Risk Screening
  * Energy and Protein Intake
  Interventions: Diagnostic Test: Quadriceps Muscle Layer Fitness; Diagnostic Test: Muscle Strength; Diagnostic Test: Acute Physiology and Chronic Health Evaluation; Diagnostic Test: Sequential Organ Failure Assessment; Diagnostic Test: Nutritional Risk Screening; Diagnostic Test: Energy and Protein Intake
- Continuous enteral feeding (Experimental): The patients randomized into this study arm will receive bolus enteral feeding.
  The study subjects will undergo the following interventions:
  * Quadriceps Muscle Layer Fitness measurement
  * Muscle Strength measurement
  * Acute Physiology and Chronic Health Evaluation
  * Sequential Organ Failure Assessment
  * Nutritional Risk Screening
  * Energy and Protein Intake
  Interventions: Diagnostic Test: Quadriceps Muscle Layer Fitness; Diagnostic Test: Muscle Strength; Diagnostic Test: Acute Physiology and Chronic Health Evaluation; Diagnostic Test: Sequential Organ Failure Assessment; Diagnostic Test: Nutritional Risk Screening; Diagnostic Test: Energy and Protein Intake

INTERVENTIONS:
Diagnostic Test: Quadriceps Muscle Layer Fitness — The QMLF examination will be performed in all study subjects, with both bolus and continuous enteral feeding.
  Other Names: QMLF
Diagnostic Test: Muscle Strength — All study subjects, with both bolus and continuous enteral feeding, will undergo measurement of the muscle strength using dynamometer.
Diagnostic Test: Acute Physiology and Chronic Health Evaluation — All study subjects, with both bolus and continuous enteral feeding, will undergo the APACHE evaluation.
  Other Names: APACHE
Diagnostic Test: Sequential Organ Failure Assessment — All study subjects, with both bolus and continuous enteral feeding, will undergo the SOFA assessment.
  Other Names: SOFA
Diagnostic Test: Nutritional Risk Screening — All study subjects, with both bolus and continuous enteral feeding, will undergo the NSR screening.
  Other Names: NSR
Diagnostic Test: Energy and Protein Intake — The amount of energy and protein supplied to the study subjects will be observed daily in all study subjects, with both bolus and continuous enteral feeding, the percentage of the planned daily intake will be analyzed.

SUMMARY:
Stress metabolisms induced by severe trauma, large abdominal surgery procedures, sepsis, etc. leads to metabolic changes, which increase energy expenditure, enhanced protein catabolism, insulin resistance. Muscle proteolysis is massively stimulated. Critically ill patients pay for survival with a loss of muscles. Enteral nutrition, especially protein delivery to critically ill, is very important for optimizing their outcome. Standard enteral feeding regiments are generally based on continuous feeding, which is thought to be better tolerated by critically ill patients with easier glycaemic control by continuous infusion of insulin, translated in less glycaemic variability. But this approach is not physiological, continuous feeding does not allow protein synthesis. Optimal protein synthesis requires a pulsatile increase in branched-chain amino acids. Bolus feeding activates the entrohormonal axis (bioactive peptides, insulin), and stimulates skeletal muscle synthesis to the maximum extent. The question is, whether bolus enteral feeding in critically ill patients with limited gastrointestinal function delivers a greater amount of protein, improves nutritional parameters, with higher quadriceps muscle layer thickness (QMLT) and muscle strength.

DETAILED DESCRIPTION:
The trial has been designed in accordance with the Recommendations for Interventional Trials (SPIRIT 2013) and the Consolidated Standards for Reporting of Trials CONSORT guidelines.

Patients who meet the study inclusion criteria (severe trauma patients, surgical patients and medical patients with sepsis, with inserted nasogastric/nasoduodenal feed-ing tube) will be eligible to participate, especially patients who are mechanically ventilated. The last criterion is not a necessary precondition (a module of indirect calorimetry will be used in these patients). The necessary condition is the elimination of shock within 24 hours from the ICU admission and tolerance of trophic enteral feed-ing (20ml/hour) at for the period of at least 24 hours. Patients will be randomized in a ratio of 1:1 within 72 hours of their admission to receive bolus or continuous enteral feeding (sealed envelopes method). In both groups, the same goals of energy and protein will be observed (Day 1-2: E 15 kcal/kg/day, protein 0.8-1 g/kg/day; Day 3-4: E 20 kcal/kg/day, protein 1. 2 g/kg/day; Day ≥ 5: E 25 kcal/kg/day, protein 1.5-2 g/kg/day), according to protocol. The bolus enteral group will receive the amount of enteral nutrition in six boluses (per 60min dose), the continuous enteral group will receive the amount using a pump, within the timeframe of 6am-24pm. The need for parenteral nutrition will be determined by treating clinical staff independently to group allocation.

Demographic data collection: (weight, high, BMI) and conditions (trauma, surgical, medical patients), Acute Physiology and Chronic Health Evaluation (APACHE) Sequential Organ Failure Assessment (SOFA), Nutritional Risk Screening (NRS 2002).

Daily observations: glucose, mean glucose changes, insulin (IU/d), energy and protein intake (administered calories divided by the calculated energy expenditure and administered protein divided by calculated protein intake) - Adjusted/calculated energy and protein (%). Feeding intolerance (tolerating less than 40% of requirements via the enteral route for ≥ 3 days, diarrhea ≥ 500ml per day or five bowel actions). Mechanically ventilated patients (Resting Energy Expenditure (REE) and Respiratory Quotient (RQ) measured with indirect calorimetry) Day 1, 3, 5, 7: Nutritional parameters (serum albumin prealbumin, C-reactive protein (CRP), urine urea, N balance).

Day 1 and 7: Muscle layer thickness (QMLT by ultrasound measurement and mid-upper arm circumference) and muscle strength (dynamometer) from baseline to discharge. Outcomes of muscle strength/ultrasound and dynamometer) will be measured by an investigator blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* polytrauma
* major abdominal surgery
* sepsis
* ICU stay
* enteral feeding tube
* artificial ventilation

Exclusion Criteria:

* contraindication of enteral feeding
* infaust prognosis
* prolonged shock (more than 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in nutritional parameters - serum albumin | 7 days
  The development of the serum albumin levels in g/dL will be observed.
Change in nutritional parameters - prealbumin | 7 days
  The development of the serum albumin levels in mg/dL will be observed.
Change in inflammatory parameters - C-reactive protein (CRP) | 7 days
  The development of inflammatory parameters in mg/L will be observed.
Change in muscle mass | 7 days
  The development of muscle mass (circumference in centimetres) will be measured.
Change in muscle strength | 7 days
  The development of muscle strength (in kilograms) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Káňová, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Fetterplace K, Deane AM, Tierney A, Beach L, Knight LD, Rechnitzer T, Forsyth A, Mourtzakis M, Presneill J, MacIsaac C. Targeted full energy and protein delivery in critically ill patients: a study protocol for a pilot randomised control trial (FEED Trial). Pilot Feasibility Stud. 2018 Feb 20;4:52. doi: 10.1186/s40814-018-0249-9. eCollection 2018. PMID 29484196
- [Background] Tillquist M, Kutsogiannis DJ, Wischmeyer PE, Kummerlen C, Leung R, Stollery D, Karvellas CJ, Preiser JC, Bird N, Kozar R, Heyland DK. Bedside ultrasound is a practical and reliable measurement tool for assessing quadriceps muscle layer thickness. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):886-90. doi: 10.1177/0148607113501327. Epub 2013 Aug 26. PMID 23980134